CLINICAL TRIAL: NCT01092052
Title: A Phase I Dose-Escalation Study of NMS-1116354 in Adult Patients With Advanced/Metastatic Solid Tumors
Brief Title: Study of NMS-1116354 in Advanced/Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Discontinuation of clinical investigation with NMS-1116354
Sponsor: Nerviano Medical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDCA-354-002
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Advanced/Metastatic Solid Tumors
Keywords: Phase I study; Advanced/Metastatic Solid Tumors; Cdc7 kinase inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: NMS-1116354

INTERVENTIONS:
Drug: NMS-1116354 — Oral daily administration for 14 consecutive days followed by 7 days of rest

SUMMARY:
The purpose of this study is to evaluate the safety profile of NMS-1116354, a CDC7 kinase inhibitor, in adult patients with advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced/metastatic solid tumors, for which no alternative effective standard therapy is available
2. Maximum of 4 regimens of prior cancer therapy allowed
3. Prior radiotherapy allowed if no more than 25% of BM reserve irradiated
4. Resolution of all acute toxic effects (excluding alopecia) of any prior anticancer therapy
5. ECOG performance status (PS) 0 or 1
6. Adult (age >/= 18 and </= 80 years) patients
7. Adequate renal, liver and BM reserve
8. Capability to swallow capsules intact

Exclusion Criteria:

1. Current enrollment in another therapeutic clinical trial
2. Known brain metastases
3. Currently active second malignancy
4. Major surgery within 4 weeks prior to treatment
5. Any of the following in the past 6 months: myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis
6. Pregnancy or breast-feeding women
7. Known active infections
8. Gastrointestinal disease or other malabsorption syndromes that would impact on drug absorption
9. Adrenal insufficiency
10. Other severe acute or chronic medical or psychiatric condition that could compromise protocol objectives

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
First cycle dose-limiting toxicities (DLTs) and related maximum tolerated dose(MTD) | 3 weeks

SECONDARY OUTCOMES:
Evaluation of pharmacokinetics: plasma concentration at different times after dosing, area under the curve (AUC), maximum plasma concentration (Cmax), time of occurence of Cmax (tmax) and half-life (t½) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Soria, MD, Principal Investigator — Institut Gustave-Roussy (IGR); Stefania Crippa, Biotech D, PhD, Study Director — Nerviano Medical Sciences
Locations (1):
- Institut Gustave-Roussy (IGR), Villejuif, France